CLINICAL TRIAL: NCT05703269
Title: Hypofractionated Radiotherapy vs Single Fraction Radiosurgery for Brain Metastasis Patients on Immunotherapy (HYPOGRYPHE)
Brief Title: Comparing Single vs Multiple Dose Radiation for Cancer Patients With Brain Metastasis and Receiving Immunotherapy
Acronym: HYPOGRYPHE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00092505; 5UG1CA189824-08 (NIH); NCI-2022-10836 (Registry Identifier: Registry ID: NCI CTRP); WF-2201 (Other: Wake Forest NCORP Research Base)
Record Dates: First submitted 2023-01-18; First posted 2023-01-30 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: NSCLC; Renal Cell Carcinoma; Breast Carcinoma; Melanoma; Brain Metastases, Adult; Non-small Cell Lung Cancer; SCLC; Small-cell Lung Cancer
Keywords: Gamma Knife; Linear Accelerator; Immune Checkpoint Inhibitor (ICI) therapy; Stereotactic Radiosurgery (SRS); Fractionated Stereotactic Radiosurgery (FSRS); Stereotactic Radiosurgery (SSRS)
MeSH Terms: conditions — Carcinoma, Renal Cell; Breast Neoplasms; Melanoma; Brain Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1 to either SSRS or FSRS, using minimization randomization strategy considering 5 prognostic factors of interest: radiosurgery platform (GK vs. LINAC), timing of immunotherapy relative to radiation (ICI within 30 days of Day 1 prior to SRS or not), surgical status (any resection cavity vs. intact metastases only), predominant tumor type (Melanoma vs. all others), and prior courses of SRS for brain metastases (yes vs. no). All baseline patient-reported outcomes and neurocognitive assessments will be collected prior to randomization to minimize bias.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SSRS = single fraction stereotactic radiosurgery (Active Comparator): SSRS is an advanced radiation technique that delivers high dose precision radiation in a single dose to discrete intracranial lesions. SSRS has recently become a standard-of-care treatment for patients with 1-4 brain metastases and is also commonly used for patients with up to 15 metastases, due to improved neurocognitive outcomes compared to whole brain radiotherapy.
  Interventions: Radiation: single fraction stereotactic radiosurgery (SSRS)
- FSRS = fractionated stereotactic radiosurgery (Experimental): FSRS is an advanced radiation technique that uses a lower dose precision radiation delivered over 3 to 5 treatments given daily or every other day to intracranial lesions.
  Interventions: Radiation: fractionated stereotactic radiosurgery (FSRS)

INTERVENTIONS:
Radiation: single fraction stereotactic radiosurgery (SSRS) — SSRS is an advanced radiation technique that delivers high dose precision radiation in a single dose to discrete intracranial lesions.
  Arms: SSRS = single fraction stereotactic radiosurgery
Radiation: fractionated stereotactic radiosurgery (FSRS) — FSRS is an advanced radiation technique that uses a lower dose precision radiation delivered over 3 to 5 treatments given daily or every other day to intracranial lesions.
  Arms: FSRS = fractionated stereotactic radiosurgery

SUMMARY:
This study is designed to see if we can lower the chance of side effects from radiation in patients with breast, kidney, small cell lung cancer, non-small cell lung cancer or melanoma that has spread to the brain and who are also being treated with immunotherapy, specifically immune checkpoint inhibitor (ICI) therapy. This study will compare the usual care treatment of single fraction stereotactic radiosurgery (SSRS) given on one day versus fractionated stereotactic radiosurgery (FSRS), which is a lower dose of radiation given over a few days to determine if FSRS is better or worse at reducing side effects than usual care treatment.

DETAILED DESCRIPTION:
This study is an open-label, randomized, Phase III trial designed to ascertain whether fractionated stereotactic radiosurgery (FSRS) results in lower incidence of Grade 2 or higher adverse radiation effect (ARE) by 9 months compared to single fraction stereotactic radiosurgery (SSRS) in patients with large brain metastases who have received or will receive immune checkpoint inhibitor (ICI) targeted to the PD-1/PD-L1 axis within 30 days of stereotactic radiosurgery (SRS). Participants will be randomized 1:1 to either SSRS or FSRS, using a minimization randomization strategy considering 5 prognostic factors of interest: radiosurgery platform (gamma knife vs. LINAC), timing of immunotherapy relative to radiation (ICI within 30 days prior to Day 1 of SRS or not), surgical status (any resection cavity vs intact metastases only), predominant tumor type (Melanoma vs. all others), and prior courses of SRS for brain metastases (yes vs. no).

ELIGIBILITY:
Inclusion Criteria:

* At least one intact brain metastasis or resection cavity ≥ 2 cm in diameter or ≥ 4 cc volume.

  * Patients at initial diagnosis of brain metastases and patients with known brain metastasis treated with systemic therapy alone are eligible.
  * Patients who have previously undergone SRS for brain metastases are eligible if all MRIs and DICOM-RT files from prior SRS courses are available for upload to TRIAD and there are no lesions requiring re-irradiation. Prior SRS data upload is NOT required prior to enrollment and randomization. Both SSRS and FSRS are acceptable.
  * Lesion volume will be approximated by measuring the lesion's three perpendicular diameters on contrast-enhanced, T1-weighted MRI and the product of those diameters will be divided by 2 to estimate the lesion volume (e.g., xyz/2). Alternatively, direct volumetric measurements via slice-by-slice contouring on a treatment planning software package can be used to calculate the total tumor volume.
  * Any extent of non-CNS disease is allowed. There is no requirement for non-CNS disease to be controlled prior to study entry.
  * For patients considered to be borderline or potentially eligible by size or volume criteria, sites have the option to send in DICOM films for central review screening.
* Age ≥ 18 years at the time of enrollment.
* Total number of brain metastases (including resection cavities) ≤ 15 on diagnostic MRI; all lesions must be amenable to SSRS and FSRS as determined by the treating radiation oncologist. Treatment must take place at a facility credentialed by the Imaging and Radiation Oncology Core (IROC) for SRS and that offers both SSRS and FSRS as treatment options.
* Total gross tumor volume must be ≤ 30 cc. Lesion volume will be approximated by measuring each lesion's three perpendicular diameters on contrast-enhanced T1 MRI and the product of those diameters will be divided by 2 (V = xyz/2). Direct volumetric measurements by contouring all lesions on all visible slices on treatment planning software is also acceptable. If there is a cavity, only gross residual disease within or adjacent to the cavity is counted toward the 30 cc total volume.
* Ability to tolerate MRI brain with gadolinium-based contrast.
* Pathologically confirmed melanoma, renal cell carcinoma, non-small cell lung cancer, small cell lung cancer, or breast cancer.
* Has received, is currently receiving, or is planned to receive immune checkpoint inhibitor therapy (defined as agent targeted to PD-1/PD-L1 axis) within 30 days of the planned first day of SSRS/FSRS. Dual ICI therapy with PD-1/PD-L1 and CTLA-4 targeted agents are allowed, but patients treated with a single agent CTLA-4 targeted agent only are ineligible.

  o It is not mandatory to wait for the results of next generation sequencing (NGS) or other molecular tumor testing to determine if the patient is planned to receive ICI if the enrolling physician feels that identification of a mutation that would preclude ICI therapy (such as an EGFR mutation in a patient with NSCLC) is unlikely to be identified.
* Karnofsky Performance Status (KPS) ≥ 50. Refer to Appendix A.
* Negative serum or urine pregnancy test within 14 days of randomization for women of child-bearing potential.
* Ability to understand and the willingness to sign written informed consent.
* Patients must be able to provide informed consent.
* Must be able to speak, read and understand English or Spanish

Exclusion Criteria:

* Prior fractionated, whole, or partial brain radiation therapy. Prior fractionated SRS is acceptable.
* Prior courses of SRS for benign tumors such as meningiomas, pituitary adenomas, schwannomas may be acceptable if the treatment is > 2cm away from the site of a metastatic lesion that would be treated on this study. The study PI or a designated co-PI must review this type of case to confirm eligibility prior to enrollment.
* Prior diagnosis ARE, including pseudoprogression or radiation necrosis/radionecrosis, or previously treated lesions being actively evaluated for possible ARE or local failure such as concerning imaging findings currently being tracked with short interval MRI.
* Leptomeningeal carcinomatosis established by lumbar puncture cytology, or MRI imaging. In the absence of a clinical indication, a lumbar puncture is not required to confirm eligibility.
* A brain metastasis that is 5 mm or less from the optic chiasm or optic nerves
* Inability to tolerate brain MRI or receive gadolinium-based contrast
* Planned or prior therapy with bevacizumab (or bevacizumab biosimilar) within 30 days of the planned first day of SRS as part of a systemic therapy regimen at study enrollment.
* Serious intercurrent illness or medical condition judged by the local investigator to compromise the patient's safety, preclude safe administration of the planned protocol treatment, or would not permit the patient to be managed according to the protocol guidelines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Estimated)
Dates: Start 2023-07-11 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of a Grade 2 or higher Adverse Radiation Effect (ARE) | 9 months
  To compare the proportion of participants experiencing Grade 2 or higher Adverse Radiation Effects (ARE) within 9 months following randomization to single fraction stereotactic radiosurgery (SSRS) vs fractionated stereotactic radiosurgery (FSRS) in patients with brain metastases ≥ 2 cm in diameter or ≥ 4cc in volume treated with concurrent immune checkpoint inhibitor (ICI) therapy.

SECONDARY OUTCOMES:
Compare time to composite end point | 9 months
  To compare the time to the composite endpoint of either local failure of a metastasis treated with SRS (as defined in Section 8.2) or first Grade 2 or higher ARE between SSRS and FSRS groups.
Compare time to local failure between SSRS and FSRS groups | 9 months
  To compare time to local failure between SSRS and FSRS groups.
Compare time to neurologic death between groups | 9 months
  To compare time to neurologic death between groups.
Compare patient-reported brain tumor specific symptom burden | 9 months
  To compare patient-reported brain tumor specific symptom burden using the MD Anderson Symptom Inventory-Brain Tumor (MDASI-BT) between SRSS or FSRS groups at 9 months.

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Lesser, MD, Study Chair — Wake Forest University Health Sciences
Locations (39):
- United States (39):
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Decatur Memorial Hospital, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - HSHS Saint Elizabeth's Hospital, O'Fallon, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Mercy Hospital Springfield, Springfield, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Overlook Medical Center, Summit, New Jersey
  - Lovelace Medical Center-Saint Joseph Square, Albuquerque, New Mexico
  - Lovelace Radiation Oncology, Albuquerque, New Mexico
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Mercy Health - Perrysburg Hospital, Perrysburg, Ohio
  - Saint Elizabeth Youngstown Hospital, Youngstown, Ohio
  - Saint Joseph's/Candler - Bluffton Campus, Bluffton, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Aspirus Langlade Hospital, Antigo, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Wake Forest NCORP Research Base is committed to following the NIH Statement on Sharing Research Data (http://grants.nih.gov/grants/guide/ notice-files/NOT-OD-03-032.html). As of July 2018, the WF NCORP RB signed an agreement with NCI to contribute de-identified data and data dictionaries from clinical trials conducted through our RB to the NCI NCTN/NCORP data archive within 6 months of primary and non-primary publications of phase II/III and phase III trials to https://nctn-data-archive.nci.nih.gov/. This will become the primary means for sharing raw data, and we will adhere to the guidelines spelled out in the NCTN/NCORP Data Archive Usage Guide. De-identified data from studies not covered by the agreement (e.g., phase II and observational studies) will be made available upon request. All data files will be de-identified.
  De-identification procedures will meet the HIPAA criteria as detailed in the Code of Federal Regulations, Part 45, Section 164.514.
Time Frame: 6 months after publication for a 2 year duration
Access Criteria: upon request to NCORP@wakehealth.edu